CLINICAL TRIAL: NCT02923882
Title: Simple and Safe "100-dollar-kitchen" to Prevent Low-birth-weight in a Rural Area in Bangladesh: A Cluster Randomized Controlled Trial
Brief Title: $100Kitchen and Low-birth-weight Study in Rural Bangladesh
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PR-12087
Record Dates: First submitted 2016-10-02; First posted 2016-10-05 (Estimated); Last update posted 2022-02-11 (Actual); Status verified 2013-03

CONDITIONS: Pregnant Women; Low-Birth-Weight Infant
Keywords: Low-birth-weight; Model kitchen; Improved cookstove

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Intervention group (Experimental): In the intervention group, the pregnant women at 8-12 weeks of gestational age used biomass fuels for cooking in the '$100Kitchen and improved cookstove'.
  Interventions: Other: '$100Kitchen and improved cookstove'
- Control group (No Intervention): In the control group, the pregnant women at 8-12 weeks of gestational age used biomass fuels for cooking in the traditional cookstove.

INTERVENTIONS:
Other: '$100Kitchen and improved cookstove'
  Arms: Intervention group

SUMMARY:
Low-birth-weight (LBW) is a major adverse pregnancy outcome in resource-poor countries. About 28% of all neonatal deaths worldwide are directly attributed to LBW. Exposure to biomass fuel during cooking is associated with LBW. There is unlikely to be any significant change in the use of biomass fuels in the near future, therefore, interventions targeted to reduce the harmful effects on poor pregnancy outcomes is warranted. To address this need, the investigators proposed a locally-made inexpensive prefabricated model of the "100-dollar-kitchen"($100Kitchen) with an improved cookstove for resource-poor settings. The improved cookstove of the $100Kitchen ensure complete incineration of the biomass fuels and thus, provided safeguard to the pregnant women using these fuels. This study has been measured the impact of our '$100Kitchen and improved cookstove' intervention as to whether a pregnant woman residing in a household with a '$100Kitchen and improved cookstove' is less likely to give birth to a LBW newborn. A cluster-randomized controlled trial has been adopted in Shahjadpur sub-district in Bangladesh and 628 and 639 pregnant women at 8-12 weeks gestational age enrolled for each intervention and control area respectively and followed-up through 42-days post-delivery. Birth outcomes have been noted and the newborns have been weighted within 72-hrs of the delivery. Non-invasive maternal blood Carbon Monoxide Hemoglobin saturation (SpCO) level between the intervention and control groups have also been measured.

DETAILED DESCRIPTION:
A single-stage cluster sampling was followed. All the 'mouzas' (revenue villages) in Shahjadpur sub-district were divided into clusters so that each cluster contained a population of about 3,000. This generated 188 clusters. 104 out of 188 clusters-52 clusters for the intervention and 52 clusters for the control group - were randomly selected for the study to enroll the required 1300 pregnant women. Each cluster was then randomly allocated to either the intervention or control group using a computer generated random sequence. The random allocation sequence was generated independently by a statistician, who had no further involvement with the study. Once allocated, in each cluster all the eligible pregnant women were identified, invited, and enrolled during door-to-door visits by the project field staff. The field staff included female health workers, with the help of existing government community health workers such as family welfare assistants. A total of 628 eligible pregnant women were enrolled in the intervention clusters and a total of 639 eligible pregnant women in the control clusters. During the enrolment in the intervention clusters, a $100Kitchen with the improved cookstoves was installed at each of the 628 pregnant women's households following the verbal and written consent of the women and the household head.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women at 8 to 12 weeks gestational age

Exclusion Criteria:

* Pregnant women more than 12 weeks gestational age

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1300 (Actual)
Dates: Start 2013-04; Primary Completion 2014-02 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Proportion of low-birth-weight (LBW) among newborns between intervention and control groups | Birth outcome was measured within 72 hours of the delivery

SECONDARY OUTCOMES:
Differences of maternal blood Carbon Monoxide Hemoglobin saturation (SpCO) level between intervention and control groups | Maternal blood Carbon Monoxide Hemoglobin saturation (SpCO) level was measured during 2nd and 3rd trimester of pregnancy

REFERENCES:
- [Derived] Ahmed A, Rahman AE, Ahmed S, Rahman F, Sujan HM, Ahmmed F, Hossain AT, Sayeed A, Hossain S, Huq NL, Quaiyum MA, Reichenbach L, El Arifeen S. Effect of low-cost kitchen with improved cookstove on birthweight of neonates in Shahjadpur, Bangladesh: a cluster-randomised controlled trial. Lancet Reg Health Southeast Asia. 2024 Jan 3;25:100342. doi: 10.1016/j.lansea.2023.100342. eCollection 2024 Jun. PMID 39021478